CLINICAL TRIAL: NCT02034422
Title: Understanding the Exercise-Hypertension Paradox: Implication for Rehabilitation
Brief Title: Understanding the Exercise-Hypertension Paradox
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: O1215-W; 1IK2RX001215 (NIH)
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Results first posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2023-10

CONDITIONS: Hypertension
Keywords: Exercise
MeSH Terms: conditions — Hypertension; Motor Activity | interventions — Antioxidants; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Specific Aim #1 (Experimental): Specific Aim 1: Determine the consequences of oxidative stress on skeletal muscle afferent feedback and muscle blood flow during exercise in hypertension. Hypothesis: Afferent feedback sensitivity, determined by passive leg movement (isolation of mechanoreceptor sensitivity) and post exercise circulatory occlusion (isolation of metaboreceptor sensitivity) will be greater in hypertension leading to the exaggerated EPR. Muscle blood flow, assessed by Doppler ultrasound during multiple exercise intensities, will be impaired in hypertension leading to exercise intolerance. Reductions in oxidative stress, achieved by an oral antioxidant treatment (Vitamins C, E and alpha lipoic acid), will reduce afferent fiber sensitivity and improve muscle blood flow in hypertension. Additionally, venous endothelial cells will express elevated markers of oxidative stress providing novel evidence that the vascular endothelium contributes to the greater oxidative stress in hypertension.
  Interventions: Dietary Supplement: Oral Antioxidant
- Specific Aim #2 (Experimental): Specific Aim 2: Determine the remediable effect of combined antioxidant treatment and exercise rehabilitation in the treatment of hypertension. Hypothesis: Acute antioxidant treatment administered prior to exercise in hypertensive patients will ameliorate the exaggerated EPR resulting in a normal and safe blood pressure response to exercise-based rehabilitation. This two-pronged approach (antioxidants and exercise training) will result in a safely achieved reduction in skeletal muscle afferent feedback facilitating improved exercise tolerance, improved muscle blood flow and ultimately reduced cardiovascular risk in this population.
  Interventions: Dietary Supplement: Oral Antioxidant; Other: Exercise rehabilitation

INTERVENTIONS:
Dietary Supplement: Oral Antioxidant — Consisting of vitamins C, E and alpha lipoic acid.
Other: Exercise rehabilitation — 8 weeks of exercise rehabilitation
  Arms: Specific Aim #2

SUMMARY:
Hypertension affects 37% of the Veteran population, making it the most common medical condition treated by the VA Health Care System. Physical activity is the first line of defense in the treatment and management of hypertension. However, individuals with hypertension have impaired muscle blood flow and exhibit exaggerated increases in blood pressure during exercise (exercise pressor reflex or EPR) leading to exercise intolerance and increased risk of stroke and heart attack. The cause of these impairments is not known, but it is highly likely that free radical production and the subsequent increase in oxidative stress plays a significant role. Two aims are proposed; Aim 1 will identify the physiological consequences of elevated oxidative stress in hypertension, and Aim 2 will utilize an antioxidant treatment to ameliorate the effects of an exaggerated EPR allowing the safe performance of a clinical exercise rehabilitation program which will then, itself, attenuate the EPR and reduce hypertension.

DETAILED DESCRIPTION:
Nearly 37% of all Veterans are clinically hypertensive, making hypertension the most common medical condition in the VA Health Care System. Importantly, of the 67 million Americans diagnosed with hypertension less than half are being effectively treated for their condition. Hypertension constitutes a major risk factor for cardiovascular disease and when left untreated leads to the development of heart failure, coronary heart disease, peripheral artery disease, stroke, and renal disease. Exercise and regular physical activity are considered the cornerstones of prevention and management of hypertension. However, individuals with hypertension exhibit exercise intolerance characterized by impaired skeletal muscle blood flow and heightened afferent fiber sensitivity leading to an exaggerated or greater than normal physiologic increase in blood pressure during exercise (i.e. exercise pressor reflex or EPR). This imbalance between the beneficial effects of exercise and exercise intolerance creates an interesting paradox, the causes and consequences of which are poorly understood. The etiology of hypertension is undoubtedly complex, however a common denominator in this condition, elevated oxidative stress, may contribute to impaired muscle blood flow and heightened skeletal muscle afferent feedback leading to the exaggerated EPR. Previous work from the investigators' laboratory and others suggests that elevated oxidative stress associated with aging impairs muscle blood flow. Additionally, free radicals, the initiators of oxidative stress, can directly stimulate skeletal muscle afferent fibers leading to the exaggerated EPR. Importantly, the role of oxidative stress in regulating muscle blood flow and afferent fiber function in human hypertension has not been determined. Preliminary studies support a significant role of oxidative stress in impairing muscle blood flow and contributing to the exaggerated EPR in hypertension. With this information as context two aims are proposed that will systematically identify the consequences of elevated oxidative stress in hypertension. Specific Aim 1 will determine the consequences of oxidative stress by examining how elevated free radicals contribute to heightened skeletal muscle afferent feedback and impaired muscle blood flow during exercise in hypertension leading to the exaggerated EPR. Additionally, vascular endothelial cells collected from an antecubital vein will provide novel insight regarding the endothelium as potential source of elevated oxidative stress in hypertension. Specific Aim 2 will determine the effectiveness of combined antioxidant therapy and exercise rehabilitation in the treatment of hypertension. The overall goal of this proposal is to provide novel information regarding the role of oxidative stress as a critical regulator of cardiovascular and hemodynamic responses to exercise in hypertension. By identifying potential causes and consequences of oxidative stress, important insight will be gained facilitating the development of novel approaches and therapeutic strategies for the treatment of hypertension. Importantly, the practical applications tested in these studies (i.e. antioxidant treatment and combined exercise rehabilitation) are designed to identify and document effective countermeasures to aid in the treatment and management of hypertension allowing for the safe performance of exercise in a large number of Veterans.

ELIGIBILITY:
Inclusion Criteria:

* A total of 72 middle-aged (40 - 60 years of age) healthy and hypertensive men and women will participate in these protocols after providing written informed consent.
* The investigators aim to include a 1 to 1 ratio of females and males in each group.
* Individuals diagnosed or presenting with stage 1 and stage 2 hypertension (range 140/90 to 179/109 mmHg, according to the seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High BP) may be eligible for this study.
* Blood pressure status will be assessed in triplicate in the laboratory during the medical exam and during a 24 hour period using ambulatory blood pressure monitoring.

  * Both methods must confer hypertension for study enrollment.
* Other than hypertension, all hypertensive patients will be otherwise healthy and free of overt disease as assessed by:

  * medical history;
  * standard blood chemistries (chem. 7 panel),
  * ECG at rest;
  * limb vascular examination (ankle-brachial BP index > 0.9);
  * resting BP > 140/90 mmHg; and
  * skinfold % body fat assessment.
* Subjects will have a body mass index (BMI) between 19 and 30 and have plasma glucose concentrations < 7.0 mmol/L under fasting conditions and < 11.1 mmol/L at 120 minutes of an oral glucose tolerance test (OGTT), as defined by the American Diabetes Association.
* To reduce heterogeneity of the hypertensive subjects while maintaining a "real world" approach the following classes of drugs will be allowed;

  * diuretics,
  * angiotensin converting enzyme (ACE) inhibitors,
  * and angiotensin II receptor blockers (ARB).
* Healthy normotensive subjects will be matched to their hypertensive counterparts and will be free from overt cardiovascular disease according to the criteria described above.

Inclusion/Exclusion criteria with specific reference to the exaggerated exercise pressor reflex:

* Hypertensive subjects must exhibit a 10 mmHg or greater increase in MAP at 25% of their workrate maximum during knee extension exercise to be included in this study.
* Established criteria defining a cut off for an "exaggerated" exercise pressor reflex does not exist.
* Therefore, the investigators have set the operational definition at a 10 mmHg or greater increase in MAP during 25% of workrate maximum knee extensor exercise.
* This 10 mmHg increase in MAP was chosen as this value closely matches the investigators' preliminary data (Figure 1) and previous reports while concomitantly corresponding to an increase in BP that is at least 2 standard deviations greater than the normotensive response (i.e. 6 2 (SD) mmHg increase in MAP at 25% of their workrate maximum).
* The magnitude of the exercise-induced increase in MAP will be determined during preliminary testing.
* It should be noted that the magnitude of the pressor response is graded in relation to exercise intensity, therefore, by establishing an inclusion criterion of 10 mmHg at 25% of workrate maximum, the lowest intensity to be used in the proposed studies, the investigators have set a conservative standard for study enrollment.

Exclusion Criteria:

* Candidates demonstrating dyslipidemia based on the National Cholesterol Education Program Guidelines of plasma total cholesterol > 240 mg/dl with LDL-cholesterol > 160 mg/dl will be excluded from participation.
* Hypertensive patients receiving dual or monotherapy treatment for hypertension may be included.
* Less frequently prescribed classes of drugs for hypertension (beta blockers, aldosterone receptor blocker, centrally acting sympatholytics, calcium channel blocker, direct vasodilators, renin inhibitors, and alpha blockers) will be excluded.
* Additionally, subjects reporting a history of myocardial infarction, unstable cardiac ischemia, recent cardiac catheterization, carotid artery disease, transient ischemic attack will be excluded.
* Participants must have no orthopedic limitations that would prohibit them from knee-extensor exercise or aerobic activity including cycle ergometry or treadmill exercise.
* Due to the age requirement of the subjects women may be either pre or post-menopausal.
* All pre-menopausal women will be studied during days 1 - 7 of their menstrual cycle to standardize the influence of female hormones.
* Women taking hormone replacement therapy (HRT) currently or in the preceding year will be excluded from the proposed studies due to the direct vascular effects of HRT and the variety of regimes employed.
* Participants will be made up of primarily Veterans.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Douglas Trinity, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (1):
- VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Specific Aim #1 | Specific Aim #2
Started | 49 | 26
Completed | 49 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Specific Aim #1 | Specific Aim #2 | Total
Number analyzed (Participants) | 49 | 26 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12) | 53 (10) | 52 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 20
  Male | 35 | 20 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 45 | 22 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 103 (9) | 106 (13) | 104 (11)

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure
Description: Blood pressure with be assessed prior to the study intervention and during exercise (Aim #1). Additionally, blood pressure will be assessed following 8 weeks of exercise rehabilitation
Time Frame: Immediate to 8 weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Specific Aim #1 | Specific Aim #2
Number analyzed (Participants) | 49 | 26
mmHg
  Baseline blood Pressure | 103 (9) | 106 (13)
  Post treatment blood pressure | 94 (9) | 101 (12)

ADVERSE EVENTS:
Time Frame: During study enrollment. Up to 8 weeks or when study has been completed.
Arm/Group | Specific Aim #1 | Specific Aim #2
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/26
Other Adverse Events (participants affected / at risk) | 0/49 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT02034422/Prot_SAP_000.pdf